CLINICAL TRIAL: NCT04017910
Title: Automated 3D Ultrasound-based Surveillance of Arteriovenous Fistula Maturation for Post-operative Hemodialysis Patients
Status: Terminated | Type: Observational
Why Stopped: Conversion to IDE
Sponsor: Sonavex, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-02; 2R44HL147423-04 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Results first posted 2021-10-18 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Arteriovenous Fistula; Arteriovenous Graft
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: EchoMark/EchoSure — Each subject will have an EchoMark implanted at the time of arteriovenous fistula creation, and undergo EchoSure and duplex imaging follow-up.

SUMMARY:
This is a two stage, prospective, multi-center study to evaluate the EchoMark and EchoSure devices in patients undergoing peripheral arteriovenous fistula creation for hemodialysis access.

DETAILED DESCRIPTION:
This is Stage 1 of a 2 stage protocol, targeting to enroll 60 patients in prospective, single arm, non-randomized, multi-center observational study to record objective data in patients undergoing upper extremity arteriovenous fistula construction with autologous tissue for the purpose of eventual hemodialysis access, in whom the EchoMark is placed at the site of vascular anastomosis. Follow-up visits include EchoSure and duplex imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients presenting for upper extremity arteriovenous fistula construction with autologous tissue for the purpose of eventual hemodialysis access where the surgeon has selected EchoMark and EchoSure as the optimal method of vascular monitoring based on clinical assessment and plan
* Patient is able to sign informed consent and able to participate in all testing associated with this clinical investigation
* Women of childbearing potential have a negative pregnancy test

Exclusion Criteria:

* Age <18 years old
* Patient unable to sign informed consent
* Patient participating in another investigational device or pharmacological study
* Prisoner or patient from vulnerable populations as defined in 45 CFR 46.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing arteriovenous fistula creation for hemodialysis access
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Roanoke Vascular Access Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- EchoMark/EchoSure Stage 1: EchoMark implantation at the time of fistula creation with scheduled follow up for EchoSure imaging of the fistula maturation process.
Period: Overall Study
Arm/Group | EchoMark/EchoSure Stage 1
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There was 1 screen fail.
Arm/Group | EchoMark/EchoSure Stage 1
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 68 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Performance: Data Collection
Description: Data collection to verify accuracy
Time Frame: 24 weeks
Population: Data was not collected.
Arm/Group | EchoMark/EchoSure Stage 1
Number analyzed (Participants) | 0

2. Primary Outcome: Performance Endpoint
Description: Data collection to understand the natural history of flow physiology in AV fistulas and classify the fistula that will fail.
Time Frame: 24 Weeks
Population: Data was not collected.
Arm/Group | EchoMark/EchoSure Stage 1
Number analyzed (Participants) | 0

3. Primary Outcome: Safety Endpoint
Description: Number of Subjects with Freedom from Serious Adverse Events (SAEs) during the EchoMark implantation procedure and sub-sequent post-operative period.
Time Frame: 24 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | EchoMark/EchoSure Stage 1
Number analyzed (Participants) | 17
Participants | 16

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | EchoMark/EchoSure Stage 1
All-Cause Mortality (participants affected / at risk) | 2/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EchoMark/EchoSure Stage 1 (N=17)
Seroma / Possible Infection (Infections and infestations) | 1 (1) — Possibly Device Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EchoMark/EchoSure Stage 1 (N=17)
Edema (Surgical and medical procedures) | 3 (3) — Not Device Related
Seroma (Surgical and medical procedures) | 3 (3) — Not Device Related

LIMITATIONS AND CAVEATS:
This was designed as 2 Stage Study. Subjects were only enrolled into Stage 1 and the study has been terminated

One immunocompromised transplant subject experienced a potential local wound infection and the event was deemed to be possibly device related.

Two subjects passed away during the study. One was deemed not to be in relation to the study device. The second was deemed possibly related due to a sudden death within the thirty-day postoperative window.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04017910/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT04017910/ICF_001.pdf